CLINICAL TRIAL: NCT06345794
Title: A Phase 1, Single-Center, Open-Label, 3-Cohort, Fixed-Sequence, Drug-Drug Interaction Study To Assess The Pharmacokinetics Of LY4100511 (DC-853) When Orally Administered Alone, When Coadministered With Itraconazole, Fluconazole, Or Carbamazepine In Healthy Adult Participants
Brief Title: A Study to Assess LY4100511 (DC-853) in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: DICE Therapeutics, Inc., a wholly owned subsidiary of Eli Lilly and Company (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Organization: Eli Lilly and Company (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: DCE853103; J5C-MC-FOAG (Other: DICE Therapeutics, a wholly owned subsidiary of Eli Lilly and Company); DCE853103 (Other: DICE Therapeutics, a wholly owned subsidiary of Eli Lilly and Company)
Record Dates: First submitted 2024-03-28; First posted 2024-04-03 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Healthy
Keywords: DC-853; LY4100511
MeSH Terms: interventions — Itraconazole; Fluconazole; Carbamazepine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- LY4100511 (DC-853) + Itraconazole (Experimental): Single oral doses of LY4100511 (DC-853) with single and multiple doses of Itraconazole administered orally.
  Interventions: Drug: LY4100511 (DC-853); Drug: Itraconazole
- LY4100511 (DC-853) + Fluconazole (Experimental): Single oral doses of LY4100511 (DC-853) with single and multiple doses of fluconazole administered orally.
  Interventions: Drug: LY4100511 (DC-853); Drug: Fluconazole
- LY4100511 (DC-853) + Carbamazepine (Experimental): Single oral doses of LY4100511 (DC-853) with single and multiple doses of Carbamazepine administered orally.
  Interventions: Drug: LY4100511 (DC-853); Drug: Carbamazepine

INTERVENTIONS:
Drug: LY4100511 (DC-853) — Administered orally.
  Other Names: DC-853
Drug: Itraconazole — Administered orally.
  Arms: LY4100511 (DC-853) + Itraconazole
Drug: Fluconazole — Administered orally.
  Arms: LY4100511 (DC-853) + Fluconazole
Drug: Carbamazepine — Administered orally.
  Arms: LY4100511 (DC-853) + Carbamazepine

SUMMARY:
The main purpose of this study is to assess the effect of multiple doses of itraconazole, fluconazole, and carbamazepine on single dose pharmacokinetic of LY4100511 (DICE-853) in healthy participants. The study will also evaluate the safety and tolerability of LY4100511 (DICE-853) with itraconazole, fluconazole, and carbamazepine.

ELIGIBILITY:
Inclusion Criteria:

* Have a body mass index within the range of 18.0 to 32 kilograms per square meter (kg/m²)
* Males who agree to follow contraceptive requirements and women of not childbearing potential
* Have body weight greater than or equal to (>=) 50 Kilograms at screening.
* Must have a negative Interferon-Gamma Release Assays (IGRA) testing at screening
* Must have been stopped all the prescribed medication at least 14 days prior to admission to the clinical site
* Ability and willingness to abstain from alcohol, caffeine, and methylxanthine-containing beverages or food 2 days prior to admission to the clinical site
* Abstain from any strenuous physical exercise from 4 days prior to admission and during confinement at the clinical site

Exclusion Criteria:

* Have a history of relevant drug and/or food allergies, or sensitivity to medications used in the current study
* Females participants who are currently breastfeeding
* Have History of alcohol abuse or drug addiction
* Unable to abstain from tobacco products within the 2 days prior to admission and during confinement at the clinical site
* Have Positive screen for hepatitis B surface antigen, hepatitis C virus (HCV) antibodies, or human immunodeficiency virus (HIV) 1 and 2 antibodies
* Consumption of any nutrients known to modulate CYP450 enzymes activity
* Are immunocompromised
* Have received live vaccine(s) (including attenuated live vaccines) or Bacillus Calmette-Guérin within 28 days of screening or intend to receive them during the study
* Have had any malignancy within the past 5 years

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2024-04-03 (Actual); Primary Completion 2024-06-18 (Actual); Study Completion 2024-06-18 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK): Maximum Observed Concentration (Cmax) of LY4100511 (DC-853) | Predose up to 26 Days
PK: PK: Area Under the Concentration Versus Time Curve From Zero to Last Measurable Concentration (AUC[0-t]) of LY4100511 (DC-853) | Predose up to 26 Days
PK: Area Under the Concentration Versus Time Curve From Zero to Infinity (AUC[0-inf]) of LY4100511 (DC-853) | Predose up to 26 Days

CONTACTS AND LOCATIONS:
Overall Officials: Contact Lilly at 1-800-LillyRx (1-800-545-5979), Study Director — Eli Lilly and Company
Locations (1):
- ICON San Antonio Clinical Research Unit, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No